CLINICAL TRIAL: NCT01336881
Title: Genetics and Biology of Liver Tumorigenesis in Children
Brief Title: Biomarkers in Tissue Samples From Young Patients With Liver Cancer
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AHEP11B1; NCI-2011-02852 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AHEP11B1 (Other: Children's Oncology Group); CDR0000698720 (Other: Clinical Trials.gov)
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Childhood Hepatoblastoma; Stage I Childhood Liver Cancer; Stage II Childhood Liver Cancer; Stage III Childhood Liver Cancer; Stage IV Childhood Liver Cancer
MeSH Terms: conditions — Hepatoblastoma | interventions — Gene Expression Profiling; Microarray Analysis; Base Sequence

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived tumor tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Correlative (tissue analysis): Archived tumor tissue samples are analyzed for hepatoblastoma and other liver tumor biomarkers by microRNA array profiling and exome sequencing. Results are then compared with patients' clinical data.
  Interventions: Genetic: RNA analysis; Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: nucleic acid sequencing; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: microarray analysis
  Other Names: gene expression profiling
Genetic: nucleic acid sequencing
  Other Names: Gene Sequencing; Molecular Biology, Nucleic Acid Sequencing
Other: diagnostic laboratory biomarker analysis

SUMMARY:
This research trial is studying biomarkers in tissue samples from young patients with liver cancer. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify biomarker signatures associated with hepatoblastoma subtypes (by microRNA array profiling), and their potential correlation with liver developmental stages as well as outcome.

II. To correlate expression array data with copy number array data.

SECONDARY OBJECTIVES:

I. To carry out a focused sequencing interrogation of amplified or deleted genomic regions as well as genes in key cell pathways involved in embryonic development and/or stem cell signaling pathways for which preliminary data suggests involvement in the pathogenesis of hepatoblastoma.

II. To perform whole exome sequencing in a subset of tumors.

OUTLINE: This is a multicenter study.

Archived tumor tissue samples are analyzed for hepatoblastoma and other liver tumor biomarkers by microRNA array profiling and exome sequencing. Results are then compared with patients' clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatoblastoma or other liver cancer including the following subtypes:

  * Pure fetal histology
  * Transitional histology
  * Small cell undifferentiated histology
* Participated on the Children's Oncology Group (COG) clinical trials
* Available data and tumor samples

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young patients with liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Biomarkers associated with hepatoblastoma subtypes and cancer stages | Baseline

SECONDARY OUTCOMES:
Genes involved in embryonic development and/or stem cell signaling pathways for which preliminary data suggests involvement in the pathogenesis of hepatoblastoma | Baseline
Exome sequencing | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gail Tomlinson, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States